CLINICAL TRIAL: NCT04052607
Title: Progestin Priming Ovarian Stimulation (PPOS) Compared With Antagonist Protocol on Live Birth Rate for Freeze-all Cycles: Recruitment is Slow Due to COVID19
Brief Title: Progestin Priming Ovarian Stimulation (PPOS) Compared With Antagonist Protocol for Freeze-all Cycles
Acronym: ANTA-PPOS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID19 Pandemic effect on 2020.
Sponsor: Ibn Sina Hospital (Other Government)
Responsible Party: Principal Investigator, Muhammad Fawzy, IVF Lab Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IbnSina-PPOS
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dydrogesterone Suppression (Experimental): Dydrogesterone 30 mg on stimulation day 5 till the trigger day to prevent luteinizing hormone (LH) surge. The stimulation is with 150-300 IU FSH/HMG starting on cycle day 2 and adjusted according to the AFC and AMH.
  Interventions: Drug: LH Suppression
- Dydrogesterone Suppression with minimal stimulation (Experimental): Dydrogesterone 30 mg on stimulation day 5 till the trigger day to prevent LH surge. The stimulation is with clomifene citrate 50 mg three times daily with150 IU FSH starting on cycle day 2 and continued every other day and adjusted according to the AFC and AMH.
  Interventions: Drug: LH Suppression
- Antagonist Suppression (Active Comparator): cetrorelix acetate 0.25 started on stimulation day 6 till the trigger day to prevent LH surge. The stimulation is with150-300 IU FSH starting on cycle day 2 and continued daily and adjusted according to the AFC and AMH.
  Interventions: Drug: LH Suppression

INTERVENTIONS:
Drug: LH Suppression — Stimulation protocols

SUMMARY:
Stimulation protocols for IVF underwent several cycles of upgrading aiming to achieve reasonable outcomes with low-cost cycles. Antagonist protocols have been introduced as effective and comparable to long agonist regarding the outcomes. However, these protocols are still costly. Alternative protocols using progestin suppressions appear options for consideration.

ELIGIBILITY:
Inclusion Criteria:

1. Women age of ≥ 18 to ≤ 40;
2. BMI of ≤ 31;
3. All indication for freeze-all
4. PCOS;
5. Women who have ≥ 1 year of primary or secondary infertility;
6. Tubal factor (unilateral, bilateral obstruction or salpingectomy);
7. Fresh ejaculate sperm of any count provided they have ≥ 1% normal forms and a motile fraction;
8. Women undergoing their first ICSI cycle or following a previous successful attempt;
9. Women undergoing only frozen-thawed embryo transfer;
10. Women with > 8 mm endometrial thickness at the day of progesterone supplementation in the transfer cycle;
11. Women with no detected uterine abnormality on transvaginal ultrasound (e.g. submucosal myomas, polyps or septa).

Exclusion Criteria:

1. Unilateral oophorectomy;
2. Uterine pathology or abnormality;
3. Abnormal karyotyping for them or their male partners;
4. History of repeated abortions or implantation failure;
5. Uncontrolled diabetes;
6. Liver or renal disease;
7. History of malignancy or borderline pathology;
8. Endometriosis;
9. Plan for PGD-A;
10. Severe male factor includes surgical sperm retrieval or cryopreserved sperm.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 56 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Live Birth after first Vitrified-warmed cycle | 42 weeks of gestation
  Delivery of one or more viable infants > 20th weeks of gestation

SECONDARY OUTCOMES:
Biochemical pregnancy | 14 days after egg retrieval
  positive human chorionic Gonadotrophin (βhCG) ≥ 10 IU/L
Clinical pregnancy | within 12 weeks of gestation
  registered sacs with a heartbeat on ultrasound at 7th weeks of gestation
Ongoing pregnancy | within 24 weeks of pregnancy
  continued viable pregnancy > 20th weeks of gestation
Miscarriage | Within 20 weeks of pregnancy
  loss of pregnancy ≤ 20th weeks of gestation
Term live-birth for vitrified-warmed transfer | Within 42 weeks of gestation
  Delivery of one or more viable infants ≥37 weeks of gestation
Preterm Birth | Within 42 weeks of gestation
  delivery of one or more viable infants < 37th weeks of gestation
Very preterm birth | Within 42 weeks of gestation
  delivery of one or more viable infants < 32nd weeks of gestation
Low birth weight babies | Within 24 hours of delivery
  Babies with < 2500 gm
Congenital malformation | Within one month of delivery
  delivery of congenitally malformed babies
Still birth | Within 42 weeks of gestation
  delivery of nonviable babies > 20 weeks of gestation
Cumulative live birth | One year from randomization
  Registered viable neonates after two vitrified-warmed transfers within one year of randomization
Fertilization | Within 6 days of culture
  presence of 2 pronuclei 17±1 hr after oocyte injection
Embryo cleavage | Within 6 days of culture
  Cleaved embryos per fertilized oocyte
Top-quality embryo on day 3 | Within 6 days of culture
  (7-8 cells with appropriate-sizes blastomeres and less than 10% fragmentation by volume
Blastocyst formation on day 5 or 6 | Within 6 days of culture
  formed blastocysts per fertilized oocyte
Top-quality blastocyst on day 5 | Within 6 days of culture
  Rounded and dense inner cell mass with many trophectodermal cells creating a connected zone and a blastocoel more than 100% by volume; ≥ 311 grade per fertilized oocyte
Cryopreservation | Within 6 days of culture
  Cryopreserved embryos per fertilized oocyte
Live-birth-implantation rate | Within 42 weeks of gestation
  Number of viable neonates per number of embryos transferred
Utilized embryos | Within 6 days of culture
  Number of cryopreserved plus transferred embryos per fertilized oocyte
Top-quality utilized embryos | Within 6 days of culture
  Number of high-quality embryos transferred plus cryopreserved per fertilized oocyte
Metaphase II oocyte | Within 24 hours of oocyte retrieval
  Mature oocyte per oocyte collected

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Fawzy, Principal Investigator — Ibnsina Hospital
Locations (3):
- Egypt (3):
  - Banon Fertility Center, Asyut
  - IbnSina IVF Center, IbnSina Hospital, Sohag
  - AlRahma Hospital, Sohag

IPD SHARING:
Plan to Share IPD: No